CLINICAL TRIAL: NCT03785002
Title: Comparison of Strength and Muscle Thickness of Recreational Sports Individuals With Vegetarian or Non-vegetarian Food Standards Adequate in Proteins
Brief Title: Comparison of the Increment of Neuromuscular Parameters in Vegetarians and Non-vegetarians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69787617.0.0000.5327
Record Dates: First submitted 2018-10-27; First posted 2018-12-24 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Strength Training; Dietary Proteins; Muscle Strength; Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vegetarian (Experimental): Individuals who do not consume meat (vegetarian dietary pattern) will undergo strength training sessions and guidance on protein intake (at least 20g for breakfast, lunch, and dinner)
  Interventions: Other: Strength training; Other: Protein intake
- non vegetarian (Active Comparator): Individuals who do consume meat (non vegetarian dietary pattern) will undergo strength training sessions and guidance on protein intake (at least 20g for breakfast, lunch, and dinner)
  Interventions: Other: Strength training; Other: Protein intake

INTERVENTIONS:
Other: Strength training — 24 strength training sessions, with approximately 1 hour duration, that will occur 2x/week
Other: Protein intake — Guidance on the adequacy of protein intake (at least 20g of protein in breakfast, lunch and dinner)

SUMMARY:
A strength training session promotes increased muscle sensitivity to protein synthesis, which lasts for 24 hours after its closure. Recent studies have shown that the subsequent intake to the training session of approximately 20g or 0.24g / kg of high-quality protein in the same meal induces a plateau in this synthesis. Thus, this study aims to compare the muscular strength between vegetarian and omnivorous athletes with adequate protein intake to reach this plateau. It will recruit 64 university sportsmen who have maintained vegetarian or omnivorous diet for at least 6 months, totalizing 32 individuals per group. After signing the Term of Consent, participants will be submitted to anthropometric and body composition assessment (via DEXA), neuromuscular tests [(ie, muscle strength - 1RM, peak torque of knee extensors (JE), muscle thickness of JE and cohort analysis (ANCOVA) will be used in order to compare the results of the study, and to compare the results of the covariance analysis (ANCOVA). the levels of the neuromuscular parameters between the groups, considering the initial values of the force and the initial muscular thickness as covariables, the other parameters will be presented in the form of mean and standard deviation or median, the differences will be considered significant for values of p <0, 05. Expected to find no differences in strength and muscle thickness between vegetarians and omnivores after adequate protein intake.

ELIGIBILITY:
Inclusion Criteria:

* Be over the age of 19 and under 60;
* Have BMI <30 kg / m²;
* Be vegetarian or omnivorous for at least 6 months;
* Have not exercised regularly for at least 6 months.
* Be available to practice bodybuilding at School of Physical Education, Physiotherapy and Dance, 2x / week, for 3 months, free (times to combine).

Exclusion Criteria

* Be vegan, vegetarian lacto or vegetarian egg
* Be a carrier of chronic diseases;
* Present physical limitations or musculoskeletal problems, which contraindicate the performance of strength exercises;
* Failure to adhere to the proposed dietary modifications, relating to the adequacy of the portion of protein per meal, due to financial unfeasibility (low income condition);
* Use of protein or amino acid, caffeine or other thermogenic food supplements.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Muscle Thickness (mm) | At the14th week of study participation.
  To compare muscle thickness (mm) of the femoral quadriceps by Ultrasound, among vegetarian and omnivorous participants.

SECONDARY OUTCOMES:
Maximal strength (kg) | At the 14th week of study participation.
  To compare maximal strength (kg), using the one- repetition maximum test (1RM) for bilateral knee extension exercises. Each subject's maximal load was determined with no more than five attempts and an adequate amount of recovery time was permitted between each attempt (3-5min). Each valid repetition was considered when subjects performed full knee extension with proper technique.
Isometric peak torque (PTiso) (N.m) | At the 14th week of study participation.
  To compare knee extensors Isometric peak torque (N.m), defined as the highest value of the torque recorded during unilateral knee extension, using an isokinetic dynamometer, among vegetarian and omnivorous participants.
Body fat free mass (g) | At the 14th week of study participation
  To compare body fat free mass by Dual-energy x-ray absorptiometry (DEXA) evaluation, of omnivorous and vegetarian participants.
Body fat mass (g) | At the14th week of study participation.
  To compare body fat mass by Dual-energy x-ray absorptiometry (DEXA) evaluation, of omnivorous and vegetarian participants.
Protein intake (g) | At the 14th week of study participation.
  To compare daily protein intake (g) assessed by 24 hour reminder, applied in interview conducted by nutritionist, of omnivorous and vegetarian participants.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina G de Souza, PHD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Gabriela Luccciana Martini, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martini GL, Pinto RS, Brusco CM, Franceschetto BF, Oliveira ML, Neske R, Cadore FL, Teodoro JL, Wilhelm EN, de Souza CG. Similar body composition, muscle size, and strength adaptations to resistance training in lacto-ovo-vegetarians and non-vegetarians. Appl Physiol Nutr Metab. 2023 Jun 1;48(6):469-478. doi: 10.1139/apnm-2022-0258. Epub 2023 Mar 1. PMID 36857740